CLINICAL TRIAL: NCT04676633
Title: Phase 1 Multicenter, Open-Label, Dose Escalation Study and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-Tumor Activity of STP705 Administered Intratumorally in Cholangiocarcinoma, Hepatocellular Carcinoma or Liver Metastases in Subjects With Advanced/Metastatic or Surgically Unresectable Solid Tumors Who Are Refractory to Standard Therapy
Brief Title: Safety, Tolerability, PK, Anti-Tumor Activity of STP705 in Subjects With Advanced/Metastatic or Surgically Unresectable Solid Tumors Who Are Refractory to Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRN-705-005
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma; Liver Metastases; Cholangiocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Accelerated titration design followed by expansion to standard 3+3 design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: STP705 20 μg dose (Experimental): Intratumoral injection, administered as a single agent on Day 1,8 and 15 of a 28-day cycle. If the patient is deriving clinical benefit from the agent it may be continued and will be administered on Day 1 of each successive cycle.
  Interventions: Drug: STP705
- Cohort 2: STP705 40 μg dose (Experimental): Intratumoral injection, administered as a single agent on Day 1,8 and 15 of a 28-day cycle. If the patient is deriving clinical benefit from the agent it may be continued and will be administered on Day 1 of each successive cycle.
  Interventions: Drug: STP705
- Cohort 3: STP705 80 μg dose (Experimental): Intratumoral injection, administered as a single agent on Day 1,8 and 15 of a 28-day cycle. If the patient is deriving clinical benefit from the agent it may be continued and will be administered on Day 1 of each successive cycle.
  Interventions: Drug: STP705
- Cohort 4: STP705 160 μg dose (Experimental): Intratumoral injection, administered as a single agent on Day 1,8 and 15 of a 28-day cycle. If the patient is deriving clinical benefit from the agent it may be continued and will be administered on Day 1 of each successive cycle.
  Interventions: Drug: STP705
- Cohort 5: STP705 320 μg dose (Experimental): Intratumoral injection, administered as a single agent on Day 1,8 and 15 of a 28-day cycle. If the patient is deriving clinical benefit from the agent it may be continued and will be administered on Day 1 of each successive cycle.
  Interventions: Drug: STP705

INTERVENTIONS:
Drug: STP705 — Investigational Product
  Other Names: STP705 POWDER FOR INJECTION

SUMMARY:
This is an open label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of STP705 administered intratumorally in cholangiocarcinoma, hepatocellular carcinoma or liver metastasis in subjects with advanced/metastatic or surgically unresectable solid tumors who are refractory to standard therapy.

Goals:

1. To determine the MTD or RP2D of STP705 when administered intratumorally into cholangiocarcinoma, hepatocellular carcinoma, or liver metastasis.
2. To establish the dose of STP705 recommended for future phase 2 studies when administered intratumorally.

DETAILED DESCRIPTION:
This is an open label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of various doses of STP705 administered intratumorally in cholangiocarcinoma, hepatocellular carcinoma or liver metastasis.

The primary objective of this study is to determine the MTD or RP2D of STP705 and to establish the dose of STP705 recommended for future phase 2 studies when administered intratumorally.

A total of up to 30 patients will be enrolled in the dose escalation phase of the study. In addition, once the MTD or recommended phase 2 dose has been established, up to 20 additional patients maybe enrolled to confirm safety and explore anti-tumor activity.

Up to five dose levels will be explored (20,40,80,160,320 μg dose levels) and will depend on the number and intensity of observed toxicity. Intermediate doses maybe explored during escalation period.

It will follow an accelerated titration design, enrolling 1 patient per dose cohort and will expand to a standard 3+3 design after.

In the accelearted titration a Grade 2 SE triggers the transition to the 3+3 part of the study. The 3+3 part of the study will start at dose level 160μg.

Subjects will be evaluated for DLTs in the first cycle of treatment and graded aacording to NCI CTCAE v5. A cycle is 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically or cytologically confirmed advanced/metastatic or surgically unresectable cholangiocarcinoma, hepatocellular carcinoma, or other solid malignancy with one or more qualifying liver metastases who are refractory to standard therapy

   * Have at least one liver tumor or metastasis (≤ 5 cm in size) that is not sub-capsular and not near any major blood vessel
   * Have no more than 7 liver lesions
   * Is deemed safe for percutaneous intra-tumoral injection by local radiologist
2. Measurable disease per RECIST v 1.1 (primary or metastatic disease)
3. ECOG performance status or 0 - 1
4. Life expectancy of at least 3 months
5. Age ≥ 18 years
6. Signed, written Institutional Review Board (IRB) approved informed consent
7. A negative serum pregnancy test (for nonsterile women of child-bearing potential)
8. Baseline Q-T corrected interval (QTc) interval of ≤ 480 msec using Frederica's formula
9. Acceptable liver function:

   * Bilirubin ≤ 1.5 times upper limit of normal
   * AST (SGOT), ALT (SGPT) and Alkaline phosphatase ≤ 5 times upper limit of normal because of cancer or metastases to the liver
10. Acceptable renal function, defined as:

    o Serum creatinine ≤ 1.5 ULN or Creatinine Clearance ≥ 30 mL/minute
11. Acceptable hematologic status:

    * Hemoglobin ≥ 8 g/dL (a transfusion is allowed if Hemoglobin stays stable thereafter)
    * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
    * Platelet count ≥100,000 plt/mm3 x 109/ L (≥ 65,000 if low platelet counts are due to splenic sequestration and portal hypertension)
12. Urinalysis with no clinically significant abnormalities
13. Acceptable coagulation status with partial thromboplastin time (PTT) and International Normalized Ratio (INR) ≤1.5 times upper limit of normal
14. Subject has adequate vitamin D level, as defined by serum total 25-Hydroxyvitamin D [25(OH)D] ≥ 20 to < 60 ng/mL
15. Completion of all previous treatments (including surgery, systemic chemotherapy and radiotherapy), as well as supportive care (including transfusion of blood, blood components and granulocyte colony-stimulation factor [G-CSF] treatment) at least 3 weeks before screening (6 weeks for nitrosoureas or mitomycin C), with no signs or symptoms of acute toxicity > Grade 1 (except alopecia)
16. For men and women of child-producing potential, the use of effective contraceptive methods during the study
17. No aspirin for ≥ 5 days in advance of intra-tumoral administration, as well as discontinuation of antiplatelet and anticoagulant medications for the appropriate amount of time

Exclusion Criteria:

1. New York Heart Association Class III or IV cardiac disease, or myocardial infarction, severe unstable angina, coronary/peripheral artery bypass graft, congestive heart failure within the past 6 months
2. Known active, uncontrolled infection with HIV or hepatitis B; patients with hepatitis B allowed if on anti-viral therapy and have a viral load ≤ 500 IU; patients with a history of HIV must be on antiretroviral therapy for at least four weeks and have an HIV viral load ≤ 400 copies/mL, have CD4+ T cell counts ≥ 350 cells/uL and no history of AIDS-defining opportunistic infections within 3 months prior to treatment
3. Hepatocellular carcinoma patients with a Child Pugh score > B7
4. Had paracentesis in the last 3 months; presence of ascites must be controlled by diuretics
5. History of hepatic encephalopathy in the last 6 months
6. History of variceal bleeding in the last 6 months
7. Concomitant medications that are strong inhibitors or inducers of CYP450 enzymes that cannot be stopped or replaced during the study
8. Major surgical procedure within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study. (Note: Placement of a central venous access catheter(s) (e.g., port or similar) is not considered a major surgical procedure.)
9. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
10. Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
11. Participation in a clinical study involving administration of an investigational compound within the past 30 days prior to study entry.
12. Previous intratumoral injection within the past 30 days prior to study entry.
13. Unwillingness or inability to comply with procedures required in this protocol
14. Known allergy or hypersensitivity to the study drug(s) or one of the ingredients in the formulation
15. Existence of any surgical, medical or laboratory condition that, in the judgment of the clinical investigator, might interfere with the safety, distribution, metabolism or excretion of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 day cycle
  Recommended starting dose & schedule
Limited Dose Toxicity (LTD) | 28 day cycle
  Recommended starting dose & dose escalation

CONTACTS AND LOCATIONS:
Overall Officials: Francois Lebel, MD, Study Director — Chief Medical Officer
Locations (4):
- United States (4):
  - Honor Health, Scottsdale, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Norton Cancer Institute, Louisville, Kentucky
  - Atlantic Health System, Morristown, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided